CLINICAL TRIAL: NCT00425711
Title: An Open-Label Study of Acamprosate in DUI Court Participants
Brief Title: Study of Acamprosate in Driving Under the Influence (DUI) Court Participants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment barriers.
Sponsor: University of Oklahoma (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Warnock_Acamprosate
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Alcohol Dependence
Keywords: Acamprosate; Alcohol Dependence; Driving Under the Influence; Drug Court; DUI Court
MeSH Terms: conditions — Alcoholism; Driving Under the Influence | interventions — Acamprosate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DUI Court Participants (Experimental): Individuals enrolled in the DUI Court treatment site will be recruited for the 13 week open-label trial of acamprosate.
  Interventions: Drug: Acamprosate

INTERVENTIONS:
Drug: Acamprosate — Acamprosate 666 mg tid, or 333 tid in renal impairment, for 12 weeks
  Other Names: Campral

SUMMARY:
Acamprosate will be given to approximately 30 DUI Court participants for 3 months and outcomes will be monitored. The hypothesis is that acamprosate will be safe and well-tolerated and that subjects' craving and other symptoms related to addiction will improve over time.

DETAILED DESCRIPTION:
Purpose: The study is a 13 week open-label study of the use of acamprosate in subjects who have elected to participate in the DUI Court program in Tulsa County. Admission to the DUI Court is completely voluntary. Participants must apply for admission, undergo an initial evaluation, and receive approval by the District Attorney's office and the presiding judge. The four-phase program requires a minimum of 1 year to complete. Each phase requires counseling, mandatory random urine drug screens, mandatory daily breathalyzer tests, a nightly curfew and that the participant be gainfully employed or in school. Currently, approximately 10% of the participants are able to complete the program in the minimum 12 month requirement. The main objective of the study is to evaluate the duration of alcohol abstinence in DUI Court participants receiving acamprosate.

Design: Thirty subjects will be enrolled in the study. New DUI court participants, within 3 months of enrollment, will be invited to participate in the trial. Qualified subjects will receive, in addition to the required DUI court assessments and treatments, a physical examination, baseline safety laboratory, study drug, psychiatric evaluation, depressive and anxiety rating scales, a personality disorder questionnaire and vital signs taken at each visit. Alcohol and substance use will be assessed by self-report and validated with review of the court-ordered laboratory and breathalyzer tests.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females age 18 - 64 years of age
2. District Attorney-approved DUI Court participants within 3 months of enrollment into DUI Court
3. Currently meets DSM-IV criteria for alcohol dependence
4. Subject agrees to alcohol abstinence as a goal
5. Women must agree to use an approved method of birth control (tubal ligation, birth control pills, IUD)
6. Negative UCG (females only)
7. Treatment with an MAOI, other antidepressants, antipsychotics, anticonvulsants, mood stabilizers, or Saint John's Wort are permissible if subject has been on a stable dose for 3 months
8. Must have the ability to comprehend key components of the informed consent and provide consent
9. Current score of 15 or less on the Beck Depression Inventory II
10. Subject has undergone detoxification and is currently abstinent from alcohol

Exclusion Criteria:

1. History of allergy to acamprosate
2. Previously failed trial of acamprosate
3. Pregnancy, lactation, or unprotected intercourse during study period
4. Lifetime diagnosis of schizophrenia or schizoaffective disorder
5. Creatinine clearance <30 mL/minute. If serum creatinine is greater than 1.4 mg/dL then the Cockcroft-Gault equation will be used to estimate creatinine clearance
6. Active suicidality, a Beck Depression Inventory II suicide item score of > 2, or a Beck Depression Inventory II total score > 15
7. Any unstable medical condition which, in the opinion of the investigator, is considered clinically significant or could affect the subject's safety or ability to complete the study
8. Use of a benzodiazepine or other sedative-hypnotic agent (including kava kava or valerian), except for eszopiclone, zaleplon, or zolpidem < 3 times weekly over the last 4 weeks

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
time until relapse, i.e. any alcohol consumption | Baseline and weeks 2, 4, 8, and 12

SECONDARY OUTCOMES:
Admission to residential treatment or jail | baseline and weeks 2, 4, 8, and 12
Depressive symptoms as measured by the Beck Depression Inventory II | baseline and weeks 2, 4, 8, and 12
Anxiety symptoms as measured by the Beck Anxiety Inventory | baseline and weeks 2, 4, 8, and 12
Penn Alcohol Craving Scale scores | baseline and weeks 2, 4, 8, and 12
Obsessive Compulsive Drinking Scale scores | baseline and weeks 2, 4, 8, and 12
Adverse events | baseline and weeks 2, 4, 8, and 12
Proportion of days on which alcohol was consumed | baseline and weeks 2, 4, 8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Julia K Warnock, M.D., Ph.D., Principal Investigator — University of Oklahoma
Locations (1):
- The University of Oklahoma, Tulsa, Tulsa, Oklahoma, United States